CLINICAL TRIAL: NCT06254456
Title: End Expiratory Occlusion Test and Tidal Volume Challenge Test for Assess Fluid Responsiveness in Prone Patients
Brief Title: Fluid Responsiveness in Prone Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bhumibol Adulyadej Hospital (Other)
Responsible Party: Principal Investigator, Thanadate Sirithanasarn, Fellowship Training in Critical Care Medicine, Bhumibol Adulyadej Hospital
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: 95/66
Record Dates: First submitted 2024-01-04; First posted 2024-02-12 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Fluid Responsiveness
Keywords: Fluid responsiveness, prone, EEOT, TVC, ARDS

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prone patients (Experimental)
  Interventions: Diagnostic Test: End expiratory occlusion test

INTERVENTIONS:
Diagnostic Test: End expiratory occlusion test — Fluid responsiveness test
  Other Names: Tidal volume challenges test

SUMMARY:
To assess fluid responsiveness in prone patient

ELIGIBILITY:
Inclusion Criteria:

* patients planed to prone position for treatment

Exclusion Criteria:

* no consent
* arrhythmia
* pregnancy
* pre existing pneumothorax
* pre existing fluid overload
* cannot insert arterial or central venous catheters

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2025-05-04 (Estimated); Study Completion 2028-07-04 (Estimated)

PRIMARY OUTCOMES:
Pulse Pressure Variation | 1 year
  Detect the pulse pressure variation from cardiac output monitoring ( A- line )

IPD SHARING:
Plan to Share IPD: No